CLINICAL TRIAL: NCT02762071
Title: Liposomal Bupivacaine vs. Interscalene Nerve Block for Pain Control After Total Shoulder Arthroplasty: A Randomized Clinical Trial
Brief Title: Liposomal Bupivacaine for Pain Control After Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00063657
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Arthropathy; Shoulder Pain; Closed Fracture Proximal Humerus, Four Part
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene Nerve Block (Active Comparator): Patients in this group will receive an interscalene nerve block containing the local anesthetic ropivacaine prior to surgery. The nerve block will be administered by a fellowship-trained anesthesiologist.
  Interventions: Drug: Interscalene Nerve Block
- Liposomal Bupivacaine (Experimental): Patients in this group will receive a periarticular injection containing liposomal bupivacaine during surgery. The injection will be administered by the surgeon.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Patients in this group will receive a periarticular injection containing liposomal bupivacaine during surgery. The injection will be administered by the surgeon.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Interscalene Nerve Block — Patients in this group will receive an interscalene nerve block containing the local anesthetic ropivacaine prior to surgery. The nerve block will be administered by a fellowship-trained anesthesiologist.
  Arms: Interscalene Nerve Block

SUMMARY:
This study will compare interscalene nerve block versus liposomal bupivacaine (Exparel) for pain control after total shoulder replacements. Each method will be assessed in terms of post operative pain scores, pain medication consumption, length of stay, complications (nerve injuries, hematomas, cardiac/respiratory events) and rate of readmission due to pain. The aims of this study will be achieved through a randomized controlled trial and cost-effectiveness analysis.

DETAILED DESCRIPTION:
After the decision to proceed with shoulder replacement surgery, patients will be asked to participate in this randomized trial. Consent will be completed after explanation of each treatment group and the data to be collected. Patients will be randomized into one of the two treatment groups by simple randomization into one of two groups: Group 1 will receive interscalene nerve block and group 2 will receive liposomal bupivacaine for postoperative analgesia. Randomization will be stratified by site.

The surgeon at each site will be trained prior to enrollment on the correct way to perform Exparel injections intraoperatively. Patients in the interscalene nerve block group will be given a single shot block in the preoperative area by a fellowship-trained anesthesiologist.

The primary outcome is pain score on a visual analog scale (VAS) at 24 hours postoperatively. VAS pain scores range from 0 (no pain) to 10 (unbearable pain). Secondary outcomes are postoperative VAS pain scores at 6, 12, 18, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, and 96 hours; VAS pain score at the first postoperative visit ; intraoperative opioid consumption; postoperative opioid consumption at days 1, 2, 3, and 4; total opioid consumption at day 1 (intraoperative + postoperative day 1); duration of stay in the post-anesthesia care unit (PACU); duration of hospital stay; and VAS score for satisfaction with pain control in the hospital and at home, assessed at participants' first postoperative visit. VAS satisfaction scores range from 0 (not satisfied) to 10 (completely satisfied).

ELIGIBILITY:
Inclusion Criteria:

* Degenerative changes of the shoulder joint (documented by radiographs) in patients planning total joint replacement with one of the study's four fellowship-trained orthopaedic surgeons.
* Patients who require revision surgeries, hemiarthroplasties, or who have chronic pain issues will be included.

Exclusion Criteria:

* Allergy to liposomal bupivacaine
* Contraindications to the interscalene nerve block such as:
* Preexisting neurologic defects
* Local anesthetic allergy
* Coagulopathy
* Contralateral phrenic nerve dysfunction
* Severe chronic obstructive pulmonary disease

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srikumaran, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Columbia, Maryland
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Patients in this group will receive a periarticular injection containing liposomal bupivacaine and with local bupivacaine during surgery. The injection will be administered by the surgeon.
Period: Overall Study
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Started | 54 | 54
Completed | 54 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 24 | 41
  >=65 years | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10) | 65 (9) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 30 | 31 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 49 | 52 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 46 | 40 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score at 24 Hours Postoperatively
Description: The primary outcome was pain score on a visual analog scale (VAS) at 24 hours postoperatively. VAS pain scores range from 0 (no pain) to 10 (unbearable pain).
Time Frame: At 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
score on a scale | 5.0 (3.0) | 4.9 (2.7)

2. Secondary Outcome: Opioid Medication Consumption in Morphine Milligram Equivalents
Description: We analyzed intraoperative opioid consumption; postoperative opioid consumption at days 1, 2, 3, and 4; total opioid consumption at day 1 (intraoperative + postoperative day 1). This was measured in morphine milligram equivalents.
Time Frame: Up to 4 days postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
morphine milligram equivalents
  Total Intraoperative + Postoperative day 1 | 38 (14) | 60 (51)
  Intraoperative | 21 (11) | 25 (14)
  Postoperative day 1 | 18 (12) | 36 (48)
  Postoperative day 2 | 9 (10) | 7 (8)
  Postoperative day 3 | 3 (6) | 4 (8)
  Postoperative day 4 | 2 (6) | 2 (5)

3. Secondary Outcome: Length of Hospital Stay
Description: Duration of stay in hospital (hours) after shoulder replacement surgery.
Time Frame: At the time of discharge from hospital, Up to 4 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
hours | 39 (20) | 36 (14)

4. Secondary Outcome: Postoperative Visual Analog Scale (VAS) Pain Scores
Description: We analyzed postoperative VAS pain scores at 6, 12, 18, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96 hours and at the first postoperative visit. VAS pain scores range from 0 (no pain) to 10 (unbearable pain).
Time Frame: Up to first postoperative visit, maximum 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
score on a scale
  6 hours postoperative | 2.9 (3.1) | 5.1 (2.9)
  12 hours postoperative | 4.0 (3.1) | 4.6 (3.0)
  18 hours postoperative | 5.2 (3.4) | 4.6 (3.1)
  30 hours postoperative | 4.8 (2.9) | 4.6 (2.7)
  36 hours postoperative | 4.1 (2.9) | 5.1 (2.2)
  42 hours postoperative | 4.0 (2.8) | 4.6 (2.8)
  48 hours postoperative | 4.2 (2.8) | 4.3 (2.7)
  54 hours postoperative | 4.2 (2.7) | 4.4 (2.5)
  60 hours postoperative | 4.1 (2.6) | 3.9 (2.1)
  66 hours postoperative | 3.8 (2.6) | 3.6 (2.2)
  72 hours postoperative | 3.8 (2.6) | 3.7 (2.6)
  78 hours postoperative | 4.0 (2.4) | 4.2 (2.6)
  84 hours postoperative | 4.0 (2.7) | 4.1 (2.6)
  90 hours postoperative | 3.9 (2.5) | 4.1 (2.5)
  96 hours postoperative | 3.8 (2.4) | 4.3 (2.8)
  1st postoperative visit | 3.4 (2.6) | 4.4 (2.5)

5. Secondary Outcome: Patient Satisfaction With Pain Management
Description: Visual Analog Scale (VAS) score for satisfaction with pain control in the hospital and at home. This was assessed at subjects' first postoperative visit.VAS satisfaction scores range from 0 (not satisfied) to 10 (completely satisfied).
Time Frame: At first postoperative visit, up to 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
score on a scale
  Satisfaction with pain management in the hospital | 8.4 (2.6) | 7.8 (3.1)
  Satisfaction with pain management at home | 8.7 (1.9) | 8.1 (2.7)

6. Secondary Outcome: Length of Stay in the Post-anesthesia Care Unit (PACU)
Description: Duration of stay in the post-anesthesia care unit (minutes) after shoulder replacement surgery.
Time Frame: At the time of discharge from PACU, Up to 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
Number analyzed (Participants) | 54 | 54
minutes | 102 (53) | 139 (77)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Interscalene Nerve Block | Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT02762071/Prot_SAP_000.pdf